CLINICAL TRIAL: NCT01179009
Title: A Safe Ketamine-Based Therapy for Treatment Resistant Depression
Brief Title: Treatment Resistant Depression (Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Florida Atlantic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201202157
Record Dates: First submitted 2010-08-02; First posted 2010-08-10 (Estimated); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression | interventions — Ketamine; Clonidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketamine 100-hour infusion (Experimental): 100-hour infusion of ketamine plus a safener (clonidine)
  Interventions: Drug: Ketamine; Drug: Clonidine
- ketamine 40-minute infusion (Active Comparator): 40-minute ketamine infusion following a 100-hours +/- placebo (saline) infusion. Participants will also receive a safener (clonidine)
  Interventions: Drug: Ketamine; Drug: Clonidine; Drug: placebo

INTERVENTIONS:
Drug: Ketamine — Controlled IV ketamine infusion (0.00225mg/kg-min. [18% (0.0125 mg/kg-min.).
  Other Names: Ketalar; Ketalin; Ketalor
Drug: Clonidine — Participants will receive an approximately 5-day pretreatment of clonidine (max. dose 1mg/day divided doses) prior to and throughout the ketamine infusion.
  Other Names: Catapares
Drug: placebo — IV saline (i.e. placebo ketamine)
  Other Names: saline
  Arms: ketamine 40-minute infusion

SUMMARY:
Treatment resistant depression (TRD) is a major public health problem. Current therapeutic options for this patient population remain limited. With all available treatments, only a sub-set of those patients who achieve an antidepressant response are likely to achieve treatment-induced remission. The need for antidepressant medication that can provide both rapid and long lasting relief of TRD symptoms is widely recognized. There is new evidence that drugs that block NMDA glutamate receptors (NMDA antagonists) are promising candidates for meeting this need. Existing studies in TRD have used only a low-dose, brief infusion of ketamine that would not be expected to re-sensitize the NMDA receptor; in agreement with this theory, these prior studies have found only temporary improvements of depression. Our key hypothesis is that a higher-dose, longer-term ketamine infusion, such as that used in chronic pain studies, would provide a more robust and lasting improvement from depression.

Accordingly, we will test whether a 100-hour ketamine infusion would be more effective than the standard 40-minute ketamine infusion currently used in other TRD studies. We will randomize subjects to one of 2 arms: (1) 100-hour (+/- 4 hours) ketamine infusion plus clonidine for the entire infusion (2) 40-minute ketamine infusion (plus clonidine) following a 100+/- hour saline infusion. All subjects will receive clonidine, an alpha-2 agonist, to minimize side effects of ketamine (namely, brief/mild psychotic and cognitive symptoms).

DETAILED DESCRIPTION:
This experiment is a pilot study involving up to 20 healthy males or females between the ages of 18-65 to test whether a 100-hour ketamine infusion plus clonidine would be more effective, with longer lasting results, then the standard 40-minute ketamine infusion (plus clonidine). Each of the 2 arms, will be evaluated using a between subject, double-blind, randomized design.

1. a. Controlled up to 100-hour IV ketamine infusion b. clonidine safener PO prior to infusion
2. a. Controlled 40-minute IV ketamine infusion b. clonidine safener PO prior to infusion c. up to 100-hour(+/-)IV placebo (saline) infusion
3. a. Controlled up to 100-hour IV ketamine infusion b. clonidine safener PO prior to infusion
4. a.Controlled up to 100-hour IV ketamine infusion b. clonidine safener PO prior to infusion

In both conditions, participants will be admitted to the Washington University School of Medicine Clinical Research Unit at Barnes-Jewish Hospital for approximately 108-hours (Monday morning-Friday evening). Pulse, blood pressure, pulse-oximetry, and an electrocardiogram strip will be routinely monitored. Serial labs and clinical/safety ratings will be done pre-, during, and post-infusion, with the last assessments being used to assure that subjects have returned to their "baseline" prior to discharge from the research unit. Participants will continue to see their primary psychiatrist throughout the study.

ELIGIBILITY:
Inclusion criteria:

1. males and females aged 18-65 years;
2. Diagnostic and Statistical Manual (DSM) IV diagnosis of Major Depressive Disorder, recurrent, severe;
3. depression must be considered treatment refractory as defined by Montgomery Asberg Depression Rating Scale (MADRS) score of 22 or above which is consistent with other studies;
4. on a stable dose of permitted antidepressant medication or no medication pre-infusion;
5. not currently psychotic and no history of psychosis within the previous 12 months; psychosis reported in the distant past may not be exclusionary if brief, per PI's judgment;
6. no history of significant clinical or intolerable side effects or complications from clonidine;
7. if a female of child-bearing potential: not pregnant or breast feeding and agrees to use birth control during the time of pre-dosing and infusions; and
8. able to give informed consent.

Exclusion Criteria:

1. confirmed bipolar disorder, schizophrenia, or schizoaffective disorder;
2. current or recent substance abuse/dependence (or any lifetime recreational ketamine or PCP use);
3. any severe Axis II personality disorder or schizophrenia spectrum disorder that, in the PI's judgment, could confound diagnosis or adherence to treatment;
4. the presence of any abnormal laboratory findings or serious medical disorder or condition that may, in the judgment of the PI, confound the assessment of relevant biologic measures or diagnoses including: clinically significant organ system dysfunction; significant and uncontrolled endocrine disease, including diabetes mellitus; hypothyroidism; cardiovascular disease; coagulopathy; significant anemia; significant acute infection; glaucoma; dehydration; epilepsy; any diagnosed cardiac condition causing documented hemodynamic compromise or dysfunction of the SA or AV node; any diagnosed respiratory condition causing documented or clinically recognized hypoxia (e.g., chronic obstructive or restrictive pulmonary disease); after evaluation, anyone determined to have a potentially compromised airway that could be difficult to intubate; fever; BMI less than 14.5; or any medical condition known to interfere with cognitive performance; medication-related exclusions include memantine, or any medication that could be considered contraindicated ketamine;
5. current treatment with any medication contraindicated with ketamine or clonidine;
6. lifetime illegal use of PCP or ketamine; no clinical use of ketamine for past 3 months
7. meets DSM-IV criteria for Mental Retardation;
8. currently hospitalized;
9. acutely suicidal or homicidal (i.e., in imminent danger with plan, urges and intent to harm oneself or others) including any prior serious attempts (e.g., those requiring hospitalization) at the PI's discretion;
10. is pregnant or breast-feeding; unwilling to use birth control if female of child bearing potential
11. unable to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-06-06 (Actual); Study Completion 2015-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lenze, MD, Principal Investigator — Washington University School of Medicine; John W Newcomer, MD, Principal Investigator — Washington University School of Medicine; Nuri B Farber, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akinfiresoye L, Tizabi Y. Antidepressant effects of AMPA and ketamine combination: role of hippocampal BDNF, synapsin, and mTOR. Psychopharmacology (Berl). 2013 Nov;230(2):291-8. doi: 10.1007/s00213-013-3153-2. Epub 2013 Jun 4. PMID 23732839
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Bowdle TA, Radant AD, Cowley DS, Kharasch ED, Strassman RJ, Roy-Byrne PP. Psychedelic effects of ketamine in healthy volunteers: relationship to steady-state plasma concentrations. Anesthesiology. 1998 Jan;88(1):82-8. doi: 10.1097/00000542-199801000-00015. PMID 9447860
- [Background] Diazgranados N, Ibrahim L, Brutsche NE, Newberg A, Kronstein P, Khalife S, Kammerer WA, Quezado Z, Luckenbaugh DA, Salvadore G, Machado-Vieira R, Manji HK, Zarate CA Jr. A randomized add-on trial of an N-methyl-D-aspartate antagonist in treatment-resistant bipolar depression. Arch Gen Psychiatry. 2010 Aug;67(8):793-802. doi: 10.1001/archgenpsychiatry.2010.90. PMID 20679587
- [Background] Drevets WC, Furey ML. Replication of scopolamine's antidepressant efficacy in major depressive disorder: a randomized, placebo-controlled clinical trial. Biol Psychiatry. 2010 Mar 1;67(5):432-8. doi: 10.1016/j.biopsych.2009.11.021. Epub 2010 Jan 15. PMID 20074703
- [Background] Duman RS, Aghajanian GK. Synaptic dysfunction in depression: potential therapeutic targets. Science. 2012 Oct 5;338(6103):68-72. doi: 10.1126/science.1222939. PMID 23042884
- [Background] Dwyer JM, Duman RS. Activation of mammalian target of rapamycin and synaptogenesis: role in the actions of rapid-acting antidepressants. Biol Psychiatry. 2013 Jun 15;73(12):1189-98. doi: 10.1016/j.biopsych.2012.11.011. Epub 2013 Jan 4. PMID 23295207
- [Background] Emnett CM, Eisenman LN, Taylor AM, Izumi Y, Zorumski CF, Mennerick S. Indistinguishable synaptic pharmacodynamics of the N-methyl-D-aspartate receptor channel blockers memantine and ketamine. Mol Pharmacol. 2013 Dec;84(6):935-47. doi: 10.1124/mol.113.089334. Epub 2013 Oct 7. PMID 24101301
- [Background] Farber NB. The NMDA receptor hypofunction model of psychosis. Ann N Y Acad Sci. 2003 Nov;1003:119-30. doi: 10.1196/annals.1300.008. PMID 14684440
- [Background] Farber NB, Foster J, Duhan NL, Olney JW. alpha 2 adrenergic agonists prevent MK-801 neurotoxicity. Neuropsychopharmacology. 1995 Jul;12(4):347-9. doi: 10.1016/0893-133X(95)00048-I. PMID 7576011
- [Background] Farber NB, Kim SH, Dikranian K, Jiang XP, Heinkel C. Receptor mechanisms and circuitry underlying NMDA antagonist neurotoxicity. Mol Psychiatry. 2002;7(1):32-43. doi: 10.1038/sj.mp.4000912. PMID 11803444
- [Background] Flemenbaum A, Zimmermann RL. Inter- and intra-rater reliability of the Brief Psychiatric Rating Scale. Psychol Rep. 1973 Jun;32(3):783-92. doi: 10.2466/pr0.1973.33.3.783. No abstract available. PMID 4704758
- [Background] Furey ML, Drevets WC. Antidepressant efficacy of the antimuscarinic drug scopolamine: a randomized, placebo-controlled clinical trial. Arch Gen Psychiatry. 2006 Oct;63(10):1121-9. doi: 10.1001/archpsyc.63.10.1121. PMID 17015814
- [Background] Goldberg ME, Torjman MC, Schwartzman RJ, Mager DE, Wainer IW. Enantioselective pharmacokinetics of (R)- and (S)-ketamine after a 5-day infusion in patients with complex regional pain syndrome. Chirality. 2011 Feb;23(2):138-43. doi: 10.1002/chir.20890. Epub 2010 Aug 27. PMID 20803495
- [Background] Handa F, Tanaka M, Nishikawa T, Toyooka H. Effects of oral clonidine premedication on side effects of intravenous ketamine anesthesia: a randomized, double-blind, placebo-controlled study. J Clin Anesth. 2000 Feb;12(1):19-24. doi: 10.1016/s0952-8180(99)00131-2. PMID 10773503
- [Background] Hartvig P, Valtysson J, Lindner KJ, Kristensen J, Karlsten R, Gustafsson LL, Persson J, Svensson JO, Oye I, Antoni G, et al. Central nervous system effects of subdissociative doses of (S)-ketamine are related to plasma and brain concentrations measured with positron emission tomography in healthy volunteers. Clin Pharmacol Ther. 1995 Aug;58(2):165-73. doi: 10.1016/0009-9236(95)90194-9. PMID 7648766
- [Background] Jevtovic-Todorovic V, Wozniak DF, Powell S, Nardi A, Olney JW. Clonidine potentiates the neuropathic pain-relieving action of MK-801 while preventing its neurotoxic and hyperactivity side effects. Brain Res. 1998 Jan 19;781(1-2):202-11. doi: 10.1016/s0006-8993(97)01247-x. PMID 9507131
- [Background] Lai R, Katalinic N, Glue P, Somogyi AA, Mitchell PB, Leyden J, Harper S, Loo CK. Pilot dose-response trial of i.v. ketamine in treatment-resistant depression. World J Biol Psychiatry. 2014 Sep;15(7):579-84. doi: 10.3109/15622975.2014.922697. Epub 2014 Jun 9. PMID 24910102
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Background] Li N, Lee B, Liu RJ, Banasr M, Dwyer JM, Iwata M, Li XY, Aghajanian G, Duman RS. mTOR-dependent synapse formation underlies the rapid antidepressant effects of NMDA antagonists. Science. 2010 Aug 20;329(5994):959-64. doi: 10.1126/science.1190287. PMID 20724638
- [Background] Liebrenz M, Stohler R, Borgeat A. Repeated intravenous ketamine therapy in a patient with treatment-resistant major depression. World J Biol Psychiatry. 2009;10(4 Pt 2):640-3. doi: 10.1080/15622970701420481. PMID 17853274
- [Background] Luckenbaugh DA, Niciu MJ, Ionescu DF, Nolan NM, Richards EM, Brutsche NE, Guevara S, Zarate CA. Do the dissociative side effects of ketamine mediate its antidepressant effects? J Affect Disord. 2014 Apr;159:56-61. doi: 10.1016/j.jad.2014.02.017. Epub 2014 Feb 18. PMID 24679390
- [Background] Moaddel R, Venkata SL, Tanga MJ, Bupp JE, Green CE, Iyer L, Furimsky A, Goldberg ME, Torjman MC, Wainer IW. A parallel chiral-achiral liquid chromatographic method for the determination of the stereoisomers of ketamine and ketamine metabolites in the plasma and urine of patients with complex regional pain syndrome. Talanta. 2010 Oct 15;82(5):1892-904. doi: 10.1016/j.talanta.2010.08.005. Epub 2010 Aug 13. PMID 20875593
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Morgan CJ, Mofeez A, Brandner B, Bromley L, Curran HV. Acute effects of ketamine on memory systems and psychotic symptoms in healthy volunteers. Neuropsychopharmacology. 2004 Jan;29(1):208-18. doi: 10.1038/sj.npp.1300342. PMID 14603267
- [Background] Mrazek DA, Hornberger JC, Altar CA, Degtiar I. A review of the clinical, economic, and societal burden of treatment-resistant depression: 1996-2013. Psychiatr Serv. 2014 Aug 1;65(8):977-87. doi: 10.1176/appi.ps.201300059. PMID 24789696
- [Background] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Background] Naughton M, Clarke G, O'Leary OF, Cryan JF, Dinan TG. A review of ketamine in affective disorders: current evidence of clinical efficacy, limitations of use and pre-clinical evidence on proposed mechanisms of action. J Affect Disord. 2014 Mar;156:24-35. doi: 10.1016/j.jad.2013.11.014. Epub 2013 Dec 10. PMID 24388038
- [Background] Neusy AJ, Lowenstein J. Blood pressure and blood pressure variability following withdrawal of propranolol and clonidine. J Clin Pharmacol. 1989 Jan;29(1):18-24. doi: 10.1002/j.1552-4604.1989.tb03232.x. PMID 2708545
- [Background] Newcomer JW, Farber NB, Jevtovic-Todorovic V, Selke G, Melson AK, Hershey T, Craft S, Olney JW. Ketamine-induced NMDA receptor hypofunction as a model of memory impairment and psychosis. Neuropsychopharmacology. 1999 Feb;20(2):106-18. doi: 10.1016/S0893-133X(98)00067-0. PMID 9885791
- [Background] Niesters M, Martini C, Dahan A. Ketamine for chronic pain: risks and benefits. Br J Clin Pharmacol. 2014 Feb;77(2):357-67. doi: 10.1111/bcp.12094. PMID 23432384
- [Background] Nitta R, Goyagi T, Nishikawa T. Combination of oral clonidine and intravenous low-dose ketamine reduces the consumption of postoperative patient-controlled analgesia morphine after spine surgery. Acta Anaesthesiol Taiwan. 2013 Mar;51(1):14-7. doi: 10.1016/j.aat.2013.03.003. Epub 2013 May 3. PMID 23711600
- [Background] Nurnberger JI Jr, Blehar MC, Kaufmann CA, York-Cooler C, Simpson SG, Harkavy-Friedman J, Severe JB, Malaspina D, Reich T. Diagnostic interview for genetic studies. Rationale, unique features, and training. NIMH Genetics Initiative. Arch Gen Psychiatry. 1994 Nov;51(11):849-59; discussion 863-4. doi: 10.1001/archpsyc.1994.03950110009002. PMID 7944874
- [Background] Paul R, Schaaff N, Padberg F, Moller HJ, Frodl T. Comparison of racemic ketamine and S-ketamine in treatment-resistant major depression: report of two cases. World J Biol Psychiatry. 2009;10(3):241-4. doi: 10.1080/15622970701714370. PMID 19224412
- [Background] Petersen T, Papakostas GI, Mahal Y, Guyker WM, Beaumont EC, Alpert JE, Fava M, Nierenberg AA. Psychosocial functioning in patients with treatment resistant depression. Eur Psychiatry. 2004 Jun;19(4):196-201. doi: 10.1016/j.eurpsy.2003.11.006. PMID 15196600
- [Background] Petersen T, Papakostas GI, Posternak MA, Kant A, Guyker WM, Iosifescu DV, Yeung AS, Nierenberg AA, Fava M. Empirical testing of two models for staging antidepressant treatment resistance. J Clin Psychopharmacol. 2005 Aug;25(4):336-41. doi: 10.1097/01.jcp.0000169036.40755.16. PMID 16012276
- [Background] Rasmussen KG, Lineberry TW, Galardy CW, Kung S, Lapid MI, Palmer BA, Ritter MJ, Schak KM, Sola CL, Hanson AJ, Frye MA. Serial infusions of low-dose ketamine for major depression. J Psychopharmacol. 2013 May;27(5):444-50. doi: 10.1177/0269881113478283. Epub 2013 Feb 20. PMID 23428794
- [Background] Schwartzman RJ, Alexander GM, Grothusen JR, Paylor T, Reichenberger E, Perreault M. Outpatient intravenous ketamine for the treatment of complex regional pain syndrome: a double-blind placebo controlled study. Pain. 2009 Dec 15;147(1-3):107-15. doi: 10.1016/j.pain.2009.08.015. Epub 2009 Sep 23. PMID 19783371
- [Background] Sigtermans MJ, van Hilten JJ, Bauer MCR, Arbous SM, Marinus J, Sarton EY, Dahan A. Ketamine produces effective and long-term pain relief in patients with Complex Regional Pain Syndrome Type 1. Pain. 2009 Oct;145(3):304-311. doi: 10.1016/j.pain.2009.06.023. Epub 2009 Jul 14. PMID 19604642
- [Background] Trevino K, McClintock SM, McDonald Fischer N, Vora A, Husain MM. Defining treatment-resistant depression: a comprehensive review of the literature. Ann Clin Psychiatry. 2014 Aug;26(3):222-32. PMID 25166485
- [Background] Webster LR, Walker MJ. Safety and efficacy of prolonged outpatient ketamine infusions for neuropathic pain. Am J Ther. 2006 Jul-Aug;13(4):300-5. doi: 10.1097/00045391-200607000-00004. PMID 16858163
- [Background] Williams JB, Kobak KA. Development and reliability of a structured interview guide for the Montgomery Asberg Depression Rating Scale (SIGMA). Br J Psychiatry. 2008 Jan;192(1):52-8. doi: 10.1192/bjp.bp.106.032532. PMID 18174510
- [Background] Zarate CA Jr, Brutsche N, Laje G, Luckenbaugh DA, Venkata SL, Ramamoorthy A, Moaddel R, Wainer IW. Relationship of ketamine's plasma metabolites with response, diagnosis, and side effects in major depression. Biol Psychiatry. 2012 Aug 15;72(4):331-8. doi: 10.1016/j.biopsych.2012.03.004. Epub 2012 Apr 18. PMID 22516044
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Derived] Siegel JS, Palanca BJA, Ances BM, Kharasch ED, Schweiger JA, Yingling MD, Snyder AZ, Nicol GE, Lenze EJ, Farber NB. Prolonged ketamine infusion modulates limbic connectivity and induces sustained remission of treatment-resistant depression. Psychopharmacology (Berl). 2021 Apr;238(4):1157-1169. doi: 10.1007/s00213-021-05762-6. Epub 2021 Jan 22. PMID 33483802
- [Derived] Lenze EJ, Farber NB, Kharasch E, Schweiger J, Yingling M, Olney J, Newcomer JW. Ninety-six hour ketamine infusion with co-administered clonidine for treatment-resistant depression: A pilot randomised controlled trial. World J Biol Psychiatry. 2016 Apr;17(3):230-8. doi: 10.3109/15622975.2016.1142607. Epub 2016 Feb 26. PMID 26919405

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2012-2014, participants were recruited via referrals and clinicaltrials.gov at Washington University School of Medicine in St. Louis, Missouri.
Groups:
- Ketamine 100-hour Infusion: 100-hour infusion of ketamine plus a safener (clonidine)
  Ketamine: Controlled IV ketamine infusion (0.00225mg/kg-min. [18% (0.0125 mg/kg-min.).
  Clonidine: Participants will receive an approximately 5-day pretreatment of clonidine (max. dose 1mg/day divided doses) prior to and throughout the ketamine infusion.
  Scopolamine Transdermal Product: Some participants will receive a scopolamine transdermal patch prior to and throughout their infusion/injections visits.
Period: Overall Study
Arm/Group | Ketamine 100-hour Infusion | Ketamine 40-minute Infusion
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine 100-hour Infusion | Ketamine 40-minute Infusion | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.8) | 46.6 (12.8) | 44.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Family History of Alcoholism [Count of Participants; unit: Participants]
  Yes | 6 | 4 | 10
  No | 3 | 6 | 9
  Unknown | 1 | 0 | 1
CGI - Severity of Illness [Count of Participants; unit: Participants] — The Clinical Global Improvement (Severity of Illness) is a 7-point scale where the anchors range from one to seven, where 1 equals normal and 7 equals among the most severely ill patients.
  Participants
    1 = Normal | 0 | 0 | 0
    2 = Borderline mentally ill | 0 | 0 | 0
    3 = Mildly ill | 0 | 0 | 0
    4 = Moderately ill | 0 | 1 | 1
    5 = Markedly ill | 9 | 9 | 18
    6 = Severely ill | 1 | 0 | 1
    7 = Among the most extremely ill patients | 0 | 0 | 0
Lifetime Major Depressive Episodes [Count of Participants; unit: Participants]
  Single | 3 | 5 | 8
  Recurrent | 7 | 5 | 12
Age of First Major Depressive Episode [Mean (Standard Deviation); unit: years] | 18.2 (6.1) | 22.0 (5.4) | 20.1 (6.0)
Duration of Current Episode [Mean (Standard Deviation); unit: years] | 8.7 (8.6) | 16.6 (12.8) | 12.7 (11.4)
Number of Antidepressant Trials [Mean (Full Range); unit: trials] | 18.4 [12 to 31] | 16.8 [7 to 23] | 17.6 [7 to 31]
Total MADRS Score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item scale that measures the severity of depression, with a higher score indicating a higher level of depression. The range of scores is 0 to 60.
  units on a scale | 31.9 (5.9) | 34.0 (3.8) | 33.0 (4.9)
Baseline HAM-D Score [Mean (Standard Deviation); unit: units on a scale] — The total Hamilton Depression (HAM-D) Rating Scale is a 17-item scale that provides an indication of depression. A higher score represents a more severe depression. Scores over 24 are indicative of severe depression. The minimum possible score is 0 while the maximum possible score is 52.
  units on a scale | 22.1 (5.3) | 21.6 (2.8) | 21.9 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item scale that measures the severity of depression, with a higher score indicating a higher level of depression. The range of scores is 0 to 60.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ketamine 100-hour Infusion | Ketamine 40-minute Infusion
Number analyzed (Participants) | 10 | 10
Scores on a scale | -9.0 (9.5) | -6.4 (8.7)
Statistical Analysis 1: Comparison: Ketamine 100-hour Infusion vs Ketamine 40-minute Infusion; Test type: Superiority; p = 0.53, ANOVA — The p-value above represents the interaction between the treatment group and time

2. Primary Outcome: Clinical Global Impression (CGI) Global Improvement Score.
Description: The Clinical Global Improvement is a 7-point scale where the anchors range from 1 (very much improved) to 7 (very much worse).
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine 100-hour Infusion | Ketamine 40-minute Infusion
Number analyzed (Participants) | 10 | 10
Participants
  Very much improved | 2 | 1
  Much improved | 2 | 1
  Minimally improved | 1 | 0
  No change | 5 | 5
  Minimally worse | 0 | 3
  Much worse | 0 | 0
  Very much worse | 0 | 0
Statistical Analysis 1: Comparison: Ketamine 100-hour Infusion vs Ketamine 40-minute Infusion; Test type: Superiority; p = 0.06, Ordinal regression — The p-value above comes from a model where the treatment group is used to predict the CGI improvement score

ADVERSE EVENTS:
Time Frame: Symptoms were measured 4 times daily over the course of the 4-day infusion using the Brief Psychiatric Rating Scale and the Clinical and Adverse Events Checklist. For symptoms that occurred on more than one assessment, the highest severity rating is reported.
Arm/Group | Ketamine 100-hour Infusion | Ketamine 40-minute Infusion
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine 100-hour Infusion (N=10) | Ketamine 40-minute Infusion (N=10)
Visual distortions and hallucinations (General disorders) | 7 (7) | 4 (4)
Unusual thoughts and delusions (General disorders) | 7 (7) | 5 (5)
Incoherent (General disorders) | 2 (2) | 1 (1)
Disorientation (General disorders) | 3 (3) | 2 (2)
Decreased Concentration/Memory Loss (General disorders) | 10 (10) | 10 (10)
Restlessness (General disorders) | 10 (10) | 8 (8)
Anxiety (General disorders) | 10 (10) | 10 (10)
Palpitations (General disorders) | 3 (3) | 4 (4)
Insomnia (General disorders) | 9 (9) | 8 (8)
Involuntary Movements (General disorders) | 1 (1) | 3 (3)
Headache (General disorders) | 9 (9) | 8 (8)
Dizziness (General disorders) | 9 (9) | 9 (9)
Nausea (General disorders) | 6 (6) | 7 (7)
Vomiting (General disorders) | 1 (1) | 1 (1)
Diplopia (General disorders) | 3 (3) | 4 (4)
Sedation (General disorders) | 9 (9) | 9 (9)
Nystagmus (General disorders) | 9 (9) | 6 (6)
Hypersalivation (General disorders) | 0 (0) | 2 (2)
Erythema/Rash (General disorders) | 5 (5) | 4 (4)

LIMITATIONS AND CAVEATS:
A pilot and feasibility study with limited statistical power due to a small sample size. Another limitation was the lack of a scale specifically measuring dissociative symptoms. In addition, the allowance of co-occurring antidepressant use could result in increased heterogeneity of responses unrelated to the study medication. Finally, the sample was ethnically homogeneous.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes